CLINICAL TRIAL: NCT00400595
Title: A Randomized Controlled Double Blind Study Using Mupirocin Versus Polysporin Triple for the Prevention of Catheter-related Infections in Patients Treated With Peritoneal Dialysis
Brief Title: Use of Ointments in Prevention of Catheter Related Infections in PD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Vanita Jassal, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 05-0850-AE
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: End Stage Renal Disease
Keywords: peritonitis; catheter related infection; exit site ointments; mupirocin; Polysporin Triple
MeSH Terms: conditions — Kidney Failure, Chronic; Peritonitis; Catheter-Related Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Polysporin tRIPLE ointment (topical ointment in widespread use for other skin lesions)
  Interventions: Drug: Polysporin Triple
- 2 (Active Comparator): Mupirocin
  Interventions: Drug: Mupirocin ointment

INTERVENTIONS:
Drug: Mupirocin ointment — topical ointment (already in widespread clinical use)
  Arms: 2
Drug: Polysporin Triple
  Arms: 1

SUMMARY:
Peritoneal dialysis (PD) is used for the treatment of end-stage renal disease in approximately 25% of patients requiring dialysis in Canada. The most common complication is bacterial infection or 'peritonitis'. Peritonitis causes severe acute abdominal pain and may lead to failure of peritoneal dialysis treatment, hospitalization or death, particularly if left untreated. Amongst the strategies used to prevent peritonitis, patients are instructed on the regular use of a prophylactic ointment around the point where the catheter exits from the body. At the present time most centers in Canada routinely prescribe mupirocin ointment for use at the exit site, however newer ointments have become available. One such ointment is Polysporin Triple. The aim of this study is to determine if catheter related infections can be significantly reduced by the routine application of Polysporin Triple in comparison to mupirocin ointment. A multi-centre, randomized, double blind, controlled study is proposed. Participants will be randomized to either mupirocin or Polysporin Triple and followed for 18 months or until the first catheter related infection, death or catheter removal. The difference in catheter related infection rates will be compared between the two groups. We anticipate the results of this study will allow clinicians to prescribe the ointment most likely to reduce infections. By doing so this will reduce the complication rate associated with peritoneal dialysis and, ultimately improve survival.

DETAILED DESCRIPTION:
Peritoneal dialysis (PD) is used for the treatment of end-stage renal disease in approximately 25% of patients requiring dialysis in Canada. The most common PD related complication is infective peritonitis, a syndrome of acute pain, cloudy peritoneal dialysate, and infection. Although many cases of peritonitis can be treated as an outpatient, recurrent or unresolving infections can result in fibrotic changes in the peritoneal membrane, catheter removal or patient death. Gram positive organisms are amongst the commonest causes of PD peritonitis; however, recent trends show an increasing rate of gram negative and fungal infections. Strategies to prevent peritonitis include the use of prophylactic topical mupirocin at the site where the PD catheter exits from the abdominal wall. Despite this and other innovations peritonitis is still diagnosed, on average, in one patient out of every 24 patients followed for a month. The aim of this study is to determine if the incidence of catheter related infections (exit site infection, tunnel infection or peritonitis) is significantly reduced by the routine application of Polysporin Triple in comparison to mupirocin ointment.A multi-centre randomized double blind, controlled study is proposed. Polysporin Triple will be compared against the current standard of care. All patients currently being treated with, or starting onto, peritoneal dialysis will be eligible. Participants will be randomized to one of two treatment arms (mupirocin; Polysporin Triple) and stratified according to a) centre b) vintage (incident versus prevalent), and c) type of PD (chronic ambulatory peritoneal dialysis vs. automated PD). Patients will be followed for 18 months or until the first catheter related infection, death or catheter removal due to technique failure. Catheter related infections will be strictly defined using current guidelines and categorized into exit site infections, infective peritonitis or tunnel infections.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide informed consent*
2. Age over 18 years
3. Has a peritoneal dialysis catheter in situ and

   * Is established on PD for more than 3 months (prevalent patients)
   * Is undergoing training for or has initiated PD within the last 3 months (incident patients)
4. Medically stable (as defined by primary nephrologist)
5. Regularly applying mupirocin ointment to catheter exit site

Exclusion Criteria:

1. Presence of acute renal failure
2. Catheter related infection at the time of recruitment or within the previous 3 months
3. Use of an oral or IV antibiotic at the time of randomization or within the previous 1 week.
4. Known allergy to any component of gentamicin or mupirocin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-02; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the time to first catheter related infection. | 2Yrs

SECONDARY OUTCOMES:
Removal of the catheter to prevent or halt progression of a catheter related infection | 2 yrs
Hospitalizations related to catheter related infection | 2 yrs
Death due to catheter-related infection | 2 yrs
All-cause mortality | 2yrs
Technique failure (i.e. transfer to hemodialysis) | 2yrs
Mupirocin or Polysporin Triple resistance | 2yrs

CONTACTS AND LOCATIONS:
Overall Officials: Vanita Jassal, MD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Scarborough General Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Result] McQuillan RF, Chiu E, Nessim S, Lok CE, Roscoe JM, Tam P, Jassal SV. A randomized controlled trial comparing mupirocin and polysporin triple ointments in peritoneal dialysis patients: the MP3 Study. Clin J Am Soc Nephrol. 2012 Feb;7(2):297-303. doi: 10.2215/CJN.07970811. Epub 2011 Dec 1. PMID 22134627
- [Derived] Jassal SV, Lok CE; MP3 Study Group. A randomized controlled trial comparing mupirocin versus Polysporin Triple for the prevention of catheter-related infections in peritoneal dialysis patients (the MP3 study). Perit Dial Int. 2008 Jan-Feb;28(1):67-72. PMID 18178950